CLINICAL TRIAL: NCT01633060
Title: A Phase III Randomized, Double Blind, Placebo Controlled Study of BKM120 With Fulvestrant, in Postmenopausal Women With Hormone Receptor-positive HER2-negative AI Treated, Locally Advanced or Metastatic Breast Cancer Who Progressed on or After mTOR Inhibitor Based Treatment
Brief Title: A Phase III Study of BKM120 With Fulvestrant in Patients With HR+,HER2-, AI Treated, Locally Advanced or Metastatic Breast Cancer Who Progressed on or After mTORi
Acronym: BELLE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis decided not to pursue further development of buparlisib program (assessment of moderate PFS benefit with know, but manageable, buparlisib profile).
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBKM120F2303; 2012-002571-34 (EudraCT Number)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Breast Cancer
Keywords: BKM120; fulvestrant; breast cancer; metastatic; locally advanced; AI treated; mTOR inhibitor; PI3K; PIK3CA; PTEN; HER2-; HR+
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Hereditary Sensory and Autonomic Neuropathies | interventions — Fulvestrant; NVP-BKM120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BKM120 100mg + Fulvestrant (Experimental): BKM120 100 mg per day and fulvestrant given until progression or as described in the protocol.
  Interventions: Drug: Fulvestrant; Drug: BKM120
- Placebo + Fulvestrant (Placebo Comparator): BKM120 matching placebo daily and fulvestrant given until progression or as described in the protocol.
  Interventions: Drug: Fulvestrant; Drug: BKM120 matching placebo

INTERVENTIONS:
Drug: Fulvestrant — Intramuscular fulvestrant 500 mg (Day 1 and Day 15 of Cycle 1 and Day 1 of every cycle thereafter)
Drug: BKM120 — BKM120 100 mg once daily
  Arms: BKM120 100mg + Fulvestrant
Drug: BKM120 matching placebo — BKM120 matching placebo, once daily
  Arms: Placebo + Fulvestrant

SUMMARY:
This study was a multicenter, randomized, double-blind, placebo-controlled Phase III study to determine the efficacy and safety of treatment with Buparlisib plus Fulvestrant vs. Placebo plus Fulvestrant in postmenopausal women with hormone Receptor-positive (HR-positive), human epidermal growth factor receptor 2-negative (HER2-negative), aromatase inhibitor (AI)-treated, locally advanced or metastatic breast cancer whose disease progressed on or after mammalian target of rapamycin inhibitor (mTORi)-based treatment.

Patients were randomized in 2:1 ratio to treatment with buparlisib 100 mg daily in combination with fulvestrant 500 mg or placebo daily in combination with fulvestrant 500 mg. Randomization was stratified according to visceral disease status (present or absent).

DETAILED DESCRIPTION:
Novartis decided not to pursue further development of buparlisib program. On 19 Dec 2016, Novartis notified the Investigators about this decision; accordingly the CBKM120F2303 study was terminated.

ELIGIBILITY:
Key inclusion criteria

* Female patients age 18 years or older
* Histologically and/or cytologically confirmed diagnosis of breast cancer
* Radiologic evidence of inoperable locally advanced or metastatic breast cancer
* Adequate tumor tissue for the analysis of PI3K-related biomarkers
* Human epidermal growth factor receptor-2 (HER2) negative disease, and a known positive hormone receptor status
* Postmenopausal women
* Prior treatment with aromatase inhibitors
* Evidence of progression to the combination of mTORi and endocrine therapy given as the last therapy prior to study entry
* Adequate bone marrow and organ function
* ECOG performance status ≤ 2

Key exclusion criteria

* Previous treatment with PI3K inhibitors, protein kinase B inhibitors or fulvestrant
* More than one chemotherapy line for metastatic disease
* Hypersensitivity to any of the excipients of buparlisib or fulvestrant
* Symptomatic central nervous system metastases
* Concurrent malignancy or malignancy within 3 years of study enrollment
* Certain drugs or radiation within 2-4 weeks of enrollment
* Increasing or chronic treatment (>5 days) with corticosteroids or another immunosuppressive agent
* Certain scores on an anxiety and depression mood questionnaire given at screening
* Acute viral hepatitis or a history of chronic or active hepatitis B virus or hepatitis C virus
* Active cardiac disease or a history of cardiac dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2012-10-03 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (175):
- United States (37):
  - University of South Alabama / Mitchell Cancer Institute Univ South AL, Mobile, Alabama
  - Ironwood Cancer and Research Centers SC, Chandler, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Compassionate Cancer Care Medical Group CCCMG, Fountain Valley, California
  - Los Angeles Hematology/Oncology Medical Group Onc Dept., Los Angeles, California
  - Cedars Sinai Medical Center SC-5, Los Angeles, California
  - University of California at Los Angeles UCLA SC, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - Rocky Mountain Cancer Centers SC, Denver, Colorado
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Emory University School of Medicine/Winship Cancer Institute Emory, Atlanta, Georgia
  - Moanalua Medical Center. Attn: Oncology Dept, Honolulu, Hawaii
  - Edward Hospital Edward Hospital, Naperville, Illinois
  - Crescent City Research Consortium, LLC SC, Metairie, Louisiana
  - Lsu Health Sciences Center/ Lsu School of Medicine Lsu, New Orleans, Louisiana
  - John Ochsner Heart and Vascular Institute Clinical Trials Ochsner 2, New Orleans, Louisiana
  - LSU Health Sciences Center Feist-Weiller Cancer Center, New Orleans, Louisiana
  - University of Maryland Medical Center Univ Maryland, Baltimore, Maryland
  - Mercy Medical Research Institute SC, Manchester, Missouri
  - Morristown Memorial Hospital Morristown Mem, Morristown, New Jersey
  - CINJ at Cooper University Hospital Dept of Onc, Voorhees Township, New Jersey
  - Clinical Research Alliance BKM120F2303, Lake Success, New York
  - Clinical Research Alliance, Lake Success, New York
  - Montefiore Medical Center Montefiore, The Bronx, New York
  - Northwest Cancer Specialists Compass Oncology -BKM, Portland, Oregon
  - Oregon Health and Science University SC-5, Portland, Oregon
  - University of Pittsburgh Cancer Institute Dept of Magee Women's Hospital, Pittsburgh, Pennsylvania
  - The West Clinic Dept. of the West Clinic, Memphis, Tennessee
  - Texas Oncology PA Dallas Presbyterian Hospital SC, Dallas, Texas
  - Texas Oncology Texas Oncology - Sammons, Dallas, Texas
  - Texas Oncology P A SC-Austin, Dallas, Texas
  - Texas Oncology P A Texas Oncology - Fort Worth (3, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Science Center Dept of Texas Tech, El Paso, Texas
  - The Methodist Hospital Cancer Center, Houston, Texas
  - US Oncology, P.A., Tyler, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Austria (4):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
- Bulgaria (4):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
  - Novartis Investigative Site, Vratsa
- Novartis Investigative Site, Montreal, Quebec, Canada
- Colombia (2):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, Tampere, Finland
- France (11):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Reims, Marne
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Brieuc Cédex
  - Novartis Investigative Site, Saint-Herblain Cédex
- Germany (20):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leer
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Velbert
- Greece (7):
  - Novartis Investigative Site, Marousi, Athens
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Patra - RIO, GR
  - Novartis Investigative Site, Thesaloniki, Thessaloniki
  - Novartis Investigative Site, Athens
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szolnok
- Italy (35):
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Benevento, BN
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Monserrato, CA
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Sora, FR
  - Novartis Investigative Site, Lecco, LC
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Ivrea, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Mirano, VE
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Frattamaggiore
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Netherlands (8):
  - Novartis Investigative Site, Maastricht, AZ
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Hoofddorp
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, Zwolle
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Novartis Investigative Site, Olsztyn, Poland
- South Korea (3):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (15):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Castellon, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santa Cruz de Tenerife
- Sweden (3):
  - Novartis Investigative Site, Kalmar
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (6):
  - Novartis Investigative Site, Blackburn, Lancashire
  - Novartis Investigative Site, Ipswich, Suffolk
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Di Leo A, Johnston S, Lee KS, Ciruelos E, Lonning PE, Janni W, O'Regan R, Mouret-Reynier MA, Kalev D, Egle D, Csoszi T, Bordonaro R, Decker T, Tjan-Heijnen VCG, Blau S, Schirone A, Weber D, El-Hashimy M, Dharan B, Sellami D, Bachelot T. Buparlisib plus fulvestrant in postmenopausal women with hormone-receptor-positive, HER2-negative, advanced breast cancer progressing on or after mTOR inhibition (BELLE-3): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Jan;19(1):87-100. doi: 10.1016/S1470-2045(17)30688-5. Epub 2017 Dec 7. PMID 29223745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 201 centers in 22 countries worldwide (Argentina, Austria, Belgium, Bulgaria, Canada, Colombia, Finland, France, Germany, Greece, Hungary, Italy, Republic of Korea, Lebanon, The Netherlands, Norway, Poland, Spain, Sweden, Thailand, UK and USA).
Pre-assignment Details: At least 420 patients were planned to be enrolled, randomized in a 2:1 ratio (two buparlisib, one placebo). A total of 432 patients were actually enrolled and analyzed (buparlisib arm: N=289; placebo arm: N=143). Not completed: in Randomization Phase=Randomized and not Treated; in Treatment Phase=Discontinued study treatment per Protocol.
Period: Randomization Phase
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Started (All randomized patients) | 289 (All randomized patients) | 143 (All randomized patients)
Completed (Randomized and treated) | 288 | 140
Not Completed | 1 | 3
Not completed — Protocol deviation | 1 | 2
Not completed — Technical problem | 0 | 1
Period: Treatment Phase
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Started (All patients in FAS that were treated) | 288 | 140
FAS - ctDNA PIK3CA Mutant (All patients in FAS with ctDNA sample and PIK3CA mutation) | 100 | 35
FAS - ctDNA PIK3CA Non-mutant (All patients in FAS with ctDNA sample and no PIK3CA mutation) | 132 | 81
Safety Set (SS) (At least 1 dose of study treatment and a 1 post baseline safety assessment) | 288 | 140
Pharmacokinetic Analysis Set (PAS) (At least one dose of Buparlisib and had at least 1 evaluable buparlisib concentration measurement) | 63 | 0
Completed | 0 | 0
Not Completed | 288 | 140
Not completed — Adverse Event | 24 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 16 | 7
Not completed — Progressive Disease | 210 | 120
Not completed — Protocol Deviation | 1 | 0
Not completed — Study Terminated by sponsor | 7 | 3
Not completed — Subject/guardian decision | 25 | 4
Not completed — Death | 4 | 3
Period: Post-Treatment Efficacy Follow-Up Phase
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Started (All patients who discontinued treatment and entered Post-Treatment Efficacy Follow-Up Phase) | 16 (All patients who entered Post-Treatment Efficacy Fup Phase) | 2 (All patients who entered Post-Treatment Efficacy Fup Phase)
Completed | 0 | 0
Not Completed | 16 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Progressive Disease | 10 | 1
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Subject/Guardian Decision | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 289 | 143 | 432
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full Analysis Set (FAS)
  Years | 60.5 (9.76) | 61.5 (9.23) | 60.8 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS)
  Participants
    Female | 289 | 143 | 432
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS)
  Participants
    American Indian or Alaska Native | 4 | 1 | 5
    Asian | 20 | 9 | 29
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 4 | 8
    White | 249 | 121 | 370
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Local Investigator Assessment - Full Analysis Set (FAS)
Description: Progression Free Survival (PFS) is defined as the time from date of randomization to the date of first radiologically documented progression or death due to any cause. If a patient did not progress or die at the time of the analysis data cut-off or start of new antineoplastic therapy, PFS was censored at the date of the last adequate tumor assessment before the earliest of the cut-off date or the start date of additional anti-neoplastic therapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria RECIST v1.1, as 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline and/or unequivocal progression of the non-target lesions and/or appearance of a new lesion. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm. Patients were followed up for approximately every 6 weeks after randomization.
Time Frame: Every 6 weeks after randomization up to a maximum of 4 years
Population: Full Analysis Set (FAS) based on Primary Analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Months | 3.9 [2.8 to 4.2] | 1.8 [1.5 to 2.8]
Statistical Analysis 1: Comparison: BKM120 100mg + Fulvestrant vs Placebo + Fulvestrant; Test type: Other — Comparison of progression-free survival (PFS) (based on local investigator assessment) between the two treatment groups using a stratified log-rank test at one-sided 2.5% level of significance; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 1-sided [lower limit 0.53]

2. Secondary Outcome: Overall Survival (OS) - Full Analysis Set (FAS)
Description: Overall Survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut-off, OS was censored at the date of last known date patient alive. Patients were followed up approximately every 6 weeks after randomization and every 3 months during survival follow-up.
Time Frame: Every 6 weeks after randomization up to a maximum of 5 years
Population: Full Analysis Set (FAS) based on Primary Analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Months | 21.2 [18.2 to 23.4] | 22.1 [17.3 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early)

3. Secondary Outcome: Progression Free Survival (PFS) by PIK3CA Mutational Status
Description: as for outcome 1
Time Frame: Every 6 weeks after randomization up to a maximum of 5 years
Population: Full Analysis Set (FAS) -ctDNA PIK3CA mutant, Full Analysis Set (FAS) - ctDNA PIK3CA non-mutant based on Primary Analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Months
  FAS ctDNA PIK3CA mutant: number analyzed (Participants) | 100 | 35
  FAS ctDNA PIK3CA mutant | 4.2 [2.8 to 6.7] | 1.6 [1.4 to 2.8]
  FAS ctDNA PIK3CA non-mutant: number analyzed (Participants) | 132 | 81
  FAS ctDNA PIK3CA non-mutant | 3.9 [2.8 to 4.3] | 2.7 [1.5 to 3.6]

4. Secondary Outcome: Overall Survival (OS) by PIK3CA Mutational Status
Description: Overall Survival (OS) by PIK3CA mutational status based on ctDNA is defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut-off, OS was censored at the date of last known date patient alive. Patients were followed up approximately every 6 weeks after randomization and every 3 months during survival follow-up.
Time Frame: Every 6 weeks after randomization up to a maximum of 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Months
  FAS ctDNA PIK3CA mutant: number analyzed (Participants) | 100 | 35
  FAS ctDNA PIK3CA mutant | 21.8 [14.7 to 25.8] | NA [14.5 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early)
  FAS ctDNA PIK3CA non-mutant: number analyzed (Participants) | 132 | 81
  FAS ctDNA PIK3CA non-mutant | 21.4 [17.3 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early) | 21.4 [17.3 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early)

5. Secondary Outcome: Overall Response Rate (ORR) by PIK3CA Mutational Status
Description: Overall Response Rate (ORR) is defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST 1.1. ORR was analyzed in the full population and by PIK3CA mutational status based on ctDNA. Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target/non target lesions: Complete Response (CR), disappearance of all target/non target lesions (all lymph nodes assigned as non-target lesions must be non-pathological in size (< 10 mm short axis)); Partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions ; Overall Response (OR)= CR+PR. Patients were followed up for the duration of the study and for approximately every 6 weeks after randomization.
Time Frame: Every 6 weeks after randomization up to a maximum of 5 years
Population: Full Analysis Set (FAS), Full Analysis Set (FAS) -ctDNA PIK3CA mutant, Full Analysis Set (FAS) - ctDNA PIK3CA non-mutant based on Primary Analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Percentage of Participants
  Full Analysis Set (FAS) | 7.6 [4.8 to 11.3] | 2.1 [0.4 to 6.0]
  FAS ctDNA PIK3CA mutant: number analyzed (Participants) | 100 | 35
  FAS ctDNA PIK3CA mutant | 10.0 [4.9 to 17.6] | 0 [0.0 to 10.0]
  FAS ctDNA PIK3CA non-mutant: number analyzed (Participants) | 132 | 81
  FAS ctDNA PIK3CA non-mutant | 7.6 [3.7 to 13.5] | 3.7 [0.8 to 10.4]

6. Secondary Outcome: Clinical Benefit Rate (CBR) by PIK3CA Mutational Status
Description: Clinical Benefit Rate (CBR) is defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR) or stable disease (SD) or Non-CR/non-PD lasting more than 14 or 24 weeks based on local investigator's assessment according to RECIST 1.1. CBR was analyzed in the full population and by PIK3CA mutational status based on ctDNA. Patients were followed up for the duration of the study and approximately every 6 weeks after randomization.
Time Frame: Week 14, Week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Percentage of Participants
  CBR>=14wks(FAS) | 33.2 [27.8 to 39.0] | 20.3 [14.0 to 27.8]
  CBR>=24wks(FAS) | 24.6 [19.7 to 29.9] | 15.4 [9.9 to 22.4]
  CBR>=14wks(FAS ctDNA PIK3CA mutant): number analyzed (Participants) | 100 | 35
  CBR>=14wks(FAS ctDNA PIK3CA mutant) | 38.0 [28.5 to 48.3] | 14.3 [4.8 to 30.3]
  CBR>=24wks(FAS ctDNA PIK3CA mutant): number analyzed (Participants) | 100 | 35
  CBR>=24wks(FAS ctDNA PIK3CA mutant) | 30.0 [21.2 to 40.0] | 11.4 [3.2 to 26.7]
  CBR>=14wks(FAS ctDNA PIK3CA non-mutant): number analyzed (Participants) | 132 | 81
  CBR>=14wks(FAS ctDNA PIK3CA non-mutant) | 36.4 [28.2 to 45.2] | 21.0 [12.7 to 31.5]
  CBR>= 24wks(FAS ctDNA PIK3CA non-mutant): number analyzed (Participants) | 132 | 81
  CBR>= 24wks(FAS ctDNA PIK3CA non-mutant) | 25.8 [18.5 to 34.1] | 14.8 [7.9 to 24.4]

7. Secondary Outcome: Long-term Safety and Tolerability in the Two Treatment Arms - Safety Set (SS)
Description: Analysis of frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths.
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment, up to 5 years
Population: Safety Set (SS) based on Final Analysis
Measure: Number; unit: Percentage of Participants
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 288 | 140
Percentage of Participants
  AEs | 97.9 | 92.9
  SAEs | 25.7 | 18.6
  Deaths | 42.7 | 48.6

8. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 in Combination With Fulvestrant at Cycle 1 Day 1 - Pharmacokinetic Analysis Set (PAS)
Description: Plasma samples were collected from the first 100 BKM120-treated patients on Cycle 1 Day 1 (at 1h, 2h, and 6h post-dose and a recommended 9h post-dose sample).
Time Frame: C1D1 1 hour post dose, C1D1 2 hour post dose, C1D1 6 hour post dose and C1D1 9 hour post dose
Population: Pharmacokinetic Analysis Set (PAS) based on Primary Analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | BKM120 100mg + Fulvestrant
Number analyzed (Participants) | 63
nanogram per milliliter (ng/mL)
  C1D1 - 1 hour post dose | 425.178 (149.6)
  C1D1 - 2 hour post dose | 615.441 (70.9)
  C1D1 - 6 hour post dose | 314.094 (41.9)
  C1D1 - 9 hour post dose | 302.899 (58.3)

9. Secondary Outcome: Predose Trough Concentration-time Profile of BKM120 in Combination With Fulvestrant Over Time - Pharmacokinetic Analysis Set (PAS)
Description: Pre-dose samples were collected for trough concentrations at Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1 and Cycle 4 Day 1.
Time Frame: C1D15, C2D1, C3D1 and C4D1
Population: Pharmacokinetic Analysis Set (PAS) based on Primary Analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | BKM120 100mg + Fulvestrant
Number analyzed (Participants) | 63
nanogram per milliliter (ng/mL)
  C1D15 | 939.978 (36.8)
  C2D1 | 880.074 (38.4)
  C3D1 | 777.026 (131.0)
  C4D1 | 1088.074 (27.0)

10. Secondary Outcome: Health-related Quality of Life (HRQoL):Time to 10% Definitive Deterioration in the Global Health Status/Quality of Life Per EORTC-QLQ-C30 - Full Analysis Set (FAS)
Description: The global health status/QoL scale score of the QLQ-C30 is identified as the primary PRO variable of interest. Physical Functioning (PF), Emotional Functioning (EF) and Social Functioning (SF) scale scores of the QLQ-C30. The time to definitive 10% deterioration is defined as the time from the randomization date to the date of an event, which is defined as a worsening (decrease) in score by at least 10% compared to baseline, with no later increase above this threshold observed during the course of the study or death due to any cause. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high /healthy level of functioning, a high score for the global health status / QoL represents a high QoL.
Time Frame: Baseline, Week 6 (C2D15), Week 12 (C4D1), then every 8 weeks until discontinuation (a cycle [C] = 4 weeks) up to 5 years.
Population: Full Analysis (FAS) based on Primary Analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Months
  EORTC QLQ-30 - Global QoL score | 5.3 [4.4 to 8.1] | 6.3 [3.0 to 9.9]
  EORTC QLQ-30 - PF scale score | 11.8 [8.1 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early) | 10.1 [7.5 to 14.6]
  EORTC QLQ-30 - EF scale score | 10.0 [6.2 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early) | 10.0 [4.9 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early)
  EORTC QLQ-30 - SF scale score | 10.0 [6.2 to 20.2] | 11.5 [6.4 to 14.6]

11. Secondary Outcome: Time to Definitive Deterioration of ECOG Performance Status From Baseline - Full Analysis Set (FAS)
Description: The Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. The ECOG Performance Scores has 5 grades: 0 = fully active, able to carry on all pre-disease performance without restriction, 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work, 2 = ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours, 3 = capable of only limited self-care, confined to bed or chair more than 50% of waking hours, 4 = completely disabled, cannot carry on any self-care, totally confined to bed or chair and 5 = dead. Definitive deterioration is defined as no improvement in the ECOG status following observation of the deterioration.
Time Frame: Screening, Baseline (Cycle 1 Day 1) and then at day 1 of each cycle and at the EOT visit
Population: Full Analysis (FAS) based on Primary Analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 100mg + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 289 | 143
Months | 18.3 [6.9 to NA] — NA: Not estimable (preliminary OS analyses). Final OS analyses not done due to early study termination (OS data collection stopped early) | 12.0 [6.4 to 14.2]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment (FPFT) until end of treatment exposure + 30 days safety follow-up.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- BKM120 100 mg + Fulvestrant: BKM120 100 mg per day and fulvestrant given until progression or as described in the protocol test.
- All Patients: All Patients
Arm/Group | BKM120 100 mg + Fulvestrant | Placebo + Fulvestrant | All Patients
All-Cause Mortality (participants affected / at risk) | 123/288 | 68/140 | 191/428
Serious Adverse Events (participants affected / at risk) | 74/288 | 26/140 | 100/428
Other Adverse Events (participants affected / at risk) | 271/288 | 113/140 | 384/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 100 mg + Fulvestrant (N=288) | Placebo + Fulvestrant (N=140) | All Patients (N=428)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 1
Intracardiac mass (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Amaurosis (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 1
Eyelid ptosis (Eye disorders) | 0 | 1 | 1
Optic atrophy (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 5
Asthenia (General disorders) | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 1
Facial pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 2
General physical health deterioration (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1
Infective thrombosis (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 0 | 4
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Electric injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 6
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 2 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Horner's syndrome (Nervous system disorders) | 1 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1
Resting tremor (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 2 | 0 | 2
Syncope (Nervous system disorders) | 2 | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Vith nerve paralysis (Nervous system disorders) | 1 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 4 | 1 | 5
Disorientation (Psychiatric disorders) | 2 | 0 | 2
Mania (Psychiatric disorders) | 1 | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 3 | 0 | 3
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Homicide (Social circumstances) | 1 | 0 | 1
Circulatory collapse (Vascular disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 100 mg + Fulvestrant (N=288) | Placebo + Fulvestrant (N=140) | All Patients (N=428)
Abdominal pain (Gastrointestinal disorders) | 16 | 6 | 22
Abdominal pain upper (Gastrointestinal disorders) | 23 | 4 | 27
Constipation (Gastrointestinal disorders) | 29 | 13 | 42
Diarrhoea (Gastrointestinal disorders) | 76 | 13 | 89
Dry mouth (Gastrointestinal disorders) | 23 | 5 | 28
Dyspepsia (Gastrointestinal disorders) | 29 | 2 | 31
Nausea (Gastrointestinal disorders) | 100 | 24 | 124
Stomatitis (Gastrointestinal disorders) | 32 | 6 | 38
Vomiting (Gastrointestinal disorders) | 27 | 13 | 40
Asthenia (General disorders) | 52 | 15 | 67
Fatigue (General disorders) | 69 | 25 | 94
Oedema peripheral (General disorders) | 18 | 2 | 20
Pyrexia (General disorders) | 20 | 8 | 28
Urinary tract infection (Infections and infestations) | 15 | 3 | 18
Alanine aminotransferase increased (Investigations) | 113 | 10 | 123
Aspartate aminotransferase increased (Investigations) | 108 | 14 | 122
Gamma-glutamyltransferase increased (Investigations) | 26 | 5 | 31
Weight decreased (Investigations) | 27 | 7 | 34
Decreased appetite (Metabolism and nutrition disorders) | 47 | 9 | 56
Hyperglycaemia (Metabolism and nutrition disorders) | 104 | 4 | 108
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 12 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 11 | 38
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 11 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 5 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 10 | 29
Dizziness (Nervous system disorders) | 35 | 10 | 45
Dysgeusia (Nervous system disorders) | 19 | 4 | 23
Headache (Nervous system disorders) | 27 | 15 | 42
Tremor (Nervous system disorders) | 18 | 0 | 18
Anxiety (Psychiatric disorders) | 51 | 15 | 66
Depression (Psychiatric disorders) | 60 | 11 | 71
Insomnia (Psychiatric disorders) | 26 | 11 | 37
Mood altered (Psychiatric disorders) | 15 | 2 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 9 | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 12 | 34
Dry skin (Skin and subcutaneous tissue disorders) | 22 | 3 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 4 | 29
Rash (Skin and subcutaneous tissue disorders) | 37 | 3 | 40
Hot flush (Vascular disorders) | 10 | 11 | 21
Hypertension (Vascular disorders) | 33 | 8 | 41

LIMITATIONS AND CAVEATS:
The primary efficacy analysis was completed by 23May16 (primary PFS analysis cutoff date). The study was later terminated and the final safety analysis was conducted up to 08Sep17. One CRF was collecting on 21Sep2017 for survival follow up (LPLV).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.